CLINICAL TRIAL: NCT07010666
Title: Beta-Hydroxybutyrate Ingestion and Cognition During Exercise-Heat Stress
Brief Title: BHB and Cognition During Exercise-Heat Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Shawn M. Arent, Professor and Chair of Exercise Science Department, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: Pro00139698
Record Dates: First submitted 2025-05-13; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — 3-Hydroxybutyric Acid; Carbohydrates; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Taste matched placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone Supplementation (Experimental): Participants received 25g of BHB ketone ester and 4 mg/kg of caffeine.
  Interventions: Dietary Supplement: Beta-Hydroxybutyrate; Dietary Supplement: Caffeine
- Control (Active Comparator): Participants received 25g of carbohydrate and 4 mg/kg of caffeine.
  Interventions: Dietary Supplement: Carbohydrate; Dietary Supplement: Caffeine

INTERVENTIONS:
Dietary Supplement: Beta-Hydroxybutyrate — 25 grams of BHB
  Arms: Ketone Supplementation
Dietary Supplement: Carbohydrate — 25 grams of carbohydrate
  Arms: Control
Dietary Supplement: Caffeine — 4 mg/kg of caffeine

SUMMARY:
The study investigates how consuming a ketone ester (BHB) along with caffeine impacts cognitive performance under heat stress, similar to what military personnel experience in hot environments. The extreme heat can impair brain function, affecting decision-making and performance, which is critical for Special Operations Forces (SOF). BHB provides an alternative energy source for the brain, potentially improving brain blood flow and cognition, particularly during "stressful" situations. By comparing ketone and carbohydrate intake with caffeine, this study aims to find better ways to maintain mental sharpness during stressful conditions. The results could help enhance the safety and effectiveness of military operations.

DETAILED DESCRIPTION:
This study aims to examine the effects of ingestion of 25g of BHB ketone ester and 4 mg/kg of caffeine on cognitive performance during exercise-heat induced hyperthermia when compared to carbohydrate combined with the same dosage of caffeine. This will be the first study to investigate the effects of ketone ester ingestion on cognition during exercise-heat induced hyperthermia in endurance-trained adults. Further, this study has the potential to impact the safety and mission success of SOF by improving cognitive performance when making critical decisions in a physiologically compromised state.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and female participants who are between 18 and 35 years of age (inclusive).
2. Are in good general health (no active or uncontrolled diseases or conditions) and can ingest the assigned amount of fluid at each visit.
3. Have a body mass index (BMI) between 17.0 and 29.9 kg/m2 (inclusive).
4. Exercise regularly as per physical activity guidelines for Americans3 [structured exercise for a minimum of 150 cumulative minutes per week (low end) to 500 cumulative minutes of exercise per week (high-end)] and willing to maintain the same level of physical activity throughout the study period.
5. Can maintain their exercise status at the beginning of the study throughout the study period.
6. Can achieve a peak oxygen consumption at screening that is at least 55 ml/kg/min.
7. Have normal or acceptable to the investigator vital signs (BP and HR) at screening.
8. Able to agree to the requirements and restrictions of this study, willing to give voluntary consent, able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Female participants who are lactating, pregnant or planning to become pregnant during the study.
2. Carry a diagnosis of diabetes.
3. Weigh less than or equal to 80 pounds at any visits.
4. Answer "yes" to any of the questions asked on the screening questionnaire.
5. Have a history of a diagnosis of celiac disease, chronic pancreatitis, steatorrhea, unstable thyroid disease, major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorder (i.e., HIV/AIDS), cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).
6. Use any dietary supplements that may impact hydration status within the 30 days prior to the baseline visit (Familiarization Trial/Visit 2). Participants must observe a 30-day washout period of no supplementation to be eligible.
7. Consume more than two standard alcoholic drinks per day.
8. Use of inhalables, smokables, or the like (e.g., cigarettes, vaporizers, water pipes, or cannabis) within 30 days prior to the first dose of the study product or for the duration of the study.
9. Have a medical condition that may impact ability to exercise or ability to ingest prescribed fluid volume.
10. Smoking tobacco products.
11. Have a history of alcohol or substance abuse in the 12 months prior to the screening visit.
12. Are cognitively impaired and/or unable to give informed consent.
13. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients, or any of the rescue medications.
14. Have a current or previous diagnosis with SARS-CoV-2 in the three months prior to screening.
15. Have had major surgery three months prior to screening or have a planned major surgery during the course of the study.
16. Have received or use test product(s) in another research study in the 28 days prior to baseline visit, or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of the current study.
17. Have any other active or unstable medical conditions or use medications, supplements, or therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Changes in Inhibitory Control by reaction time (Go/No go) | On the experimental visit days: At Baseline (0 minutes prior to the exercise protocol), 45 minutes after baseline (exercise protocol midpoint), 90 minutes after baseline (end of the exercise protocol).
  To determine if the intervention has an impact on inhibitory control by measuring reaction time to Go targets (hits).
Changes in Inhibitory Control by reaction time by errors (Go/No go) | On the experimental visit days: At Baseline (0 minutes prior to the exercise protocol), 45 minutes after baseline (exercise protocol midpoint), 90 minutes after baseline (end of the exercise protocol).
  To determine if the intervention has an impact on inhibitory control by measuring errors of commission representing incorrect responses to the target NoGo (false alarm).
Changes in Attention (Go/No go) | On the experimental visit days: At Baseline (0 minutes prior to the exercise protocol), 45 minutes after baseline (exercise protocol midpoint), 90 minutes after baseline (end of the exercise protocol).
  To determine if the device has an impact on attention by measuring errors of omission to the target Go (misses).
Changes in Object Hit and Avoid (OHA) task: Total accuracy, Target accuracy, and Non-target accuracy | On the experimental visit days: At Baseline (0 minutes prior to the exercise protocol), 45 minutes after baseline (exercise protocol midpoint), 90 minutes after baseline (end of the exercise protocol).
  To determine the effects of the intervention on rapid response execution and inhibition during complex continuous task performance, changes in total accuracy, target accuracy, and non-target accuracy in response to the intervention will be assessed.
Changes in 1-Back Task | On the experimental visit days: At Baseline (0 minutes prior to the exercise protocol), 45 minutes after baseline (exercise protocol midpoint), 90 minutes after baseline (end of the exercise protocol).
  The determine the effects of the intervention on working memory capacity.
Changes in 2-Back Task | On the experimental visit days: At Baseline (0 minutes prior to the exercise protocol), 45 minutes after baseline (exercise protocol midpoint), 90 minutes after baseline (end of the exercise protocol).
  The determine the effects of the intervention on working memory capacity.
Changes in Hopkins Verbal Learning Task | On the experimental visit days: At Baseline (0 minutes prior to the exercise protocol), 45 minutes after baseline (exercise protocol midpoint), 90 minutes after baseline (end of the exercise protocol).
  The determine the effects of the intervention on verbal learning and memory

SECONDARY OUTCOMES:
Heart Rate | Heart rate monitors will be outfitted at baseline (at the beginning of experimental visits) and heart will be measured continuously throughout experimental visit days (approximately 2 hours per day). Maximum and average heart rates will be recorded.
  Changes in heart rate across the visit
Core Body Temperature | rectal thermometers outfitted at baseline (at the beginning of experimental visits) and core temperature will be measured continuously throughout experimental visit days (approximately 2 hours per day). Maximum and average temperature will be recorded.
  Changes in core body temperature across the visit
Blood Ketone Levels | On the experimental visit days: At Baseline (0 minutes prior to the exercise protocol), 45 minutes after baseline (exercise protocol midpoint), 90 minutes after baseline (end of the exercise protocol).
  Changes in blood ketone levels across the visit
Blood Glucose Levels | On the experimental visit days: At Baseline (0 minutes prior to the exercise protocol), 45 minutes after baseline (exercise protocol midpoint), 90 minutes after baseline (end of the exercise protocol).
  Changes in blood glucose levels across the visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No